CLINICAL TRIAL: NCT05424575
Title: Modified Fraility Index: Is it a Predictor for Early Postoperative Complications
Brief Title: Modified Fraility Index in Patients Undergoing Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Sanem Cakar Turhan, Assoc. Prof., MD, Ankara University
Other Study IDs: AU I2-59-19
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Frailty Syndrome; Postoperative Complications
Keywords: arthroplasty, fraility
MeSH Terms: conditions — Frailty; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Nonfrail (Group NF): Modified fraility index was calculated in all patients. Modified fraility index < 0.27 were included to Group NF.
- Group Frail (Group F): Modified fraility index was calculated in all patients. Modified fraility index ≥ 0.27 were included to Group F.

SUMMARY:
The authors aimed to evaluate the relation between Modified Fraility Index (MFI) and postoperative complications (myocardial infarction, cardiac arrest, pulmonary embolism, septic shock, postoperative dialysis requirement, cerebrovascular event, reintubation, prolonged mechanical ventilation, surgical wound complications), duration of hospitalization, requirement for intensive care unit (ICU) admission and rehospitalization and 30th day mortality in patients undergoing arthroplasy.

DETAILED DESCRIPTION:
Fraility index is calculated according to 70 parameters which are present in national surgical quality improvement programme (NSQIP) of American College of Surgeons. This model defines fraility as a cumulative effect of individual defects depending on clinical symptoms, disease states and disabilities which provides more accurate evaluation of aging. These 70 parameters present in NSQIP database were matched with 11 variables to create a modified fraility index.

There are 11 parametres in Modified Fraility Index (MFI) (Exacerbation of chronic obstructive pulmonary disease or history of pneumonia (within last 30 days), exacerbation of congestive heart failure (within last 30 days), diabetes mellitus, dependant functional status (partially or totally dependant), history of angina, percutaneous coronary intervention or coronary bypass grefting) (within last 30 days), medically treated hypertension, acute impaired sensorium, history of peripheral vascular disease, history of myocardial infarction (within last 6 months), cerebrovascular disease with neurological deficit, cerebrovascular disease without neurological deficit or transient ischemic attack (TIA).

Presence of one of the above MFI parameters has taken 1 point. The total point that each individual achieved according to the presence of the parameters is calculated and the total score divided by 11 is defined as MFI value.

145 patients aged between 45-85 who had undergone primary or revision total knee and hip arthroplasty were included to the current prospective study. In all patients MFI was calculated.

Patients were classified as nonfrail (MFI<0,27), and frail patients (MFI≥0.27) according to MFI value.

All patients were followed up for 30 days during postoperative period. The presence of myocardial infarction, cardiac arrest, pulmonary embolism, septic shock, postoperative dialysis requirement, cerebrovascular event, reintubation, reoperation, prolonged mechanical ventilation, surgical wound complications; duration of hospitalization; requirement for intensive care unit (ICU) admission and rehospitalization and 30th day mortality were questioned.

ELIGIBILITY:
Inclusion Criteria:

patients aged between 45-85 undergoing primary or revision total knee and hip arthroplasty

Exclusion Criteria:

Emergent surgery, patients aged below 45 and above 85, patients with cognitive dysfunction

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients aged between 45-85 undergoing primary or revision total knee and hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 30 day
  myocardial infarction, cardiac arrest, pulmonary embolism, septic shock, postoperative dialysis requirement, cerebrovascular event, reintubation, prolonged mechanical ventilation, surgical wound complications, duration of hospitalization, requirement for intensive care unit (ICU) admission and rehospitalization

SECONDARY OUTCOMES:
mortality | 30 day
  30th day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sanem Cakar Turhan, Assoc. Prof., Study Chair — Ankara University Medical School Department of Anesthesiology and ICU; Leyla Alıbaylı, Specialist, Principal Investigator — Ankara University Medical School Department of Anesthesiology and ICU; Volkan Baytas, Specialist, Principal Investigator — Ankara University Medical School Department of Anesthesiology and ICU; Suheyla Karadag Erkoc, Specialist, Principal Investigator — Ankara University Medical School Department of Anesthesiology and ICU; Onat Bermede, Specialist, Principal Investigator — Ankara University Medical School Department of Anesthesiology and ICU; Hakan Kocaoglu, Assoc. Prof., Principal Investigator — Ankara University
Locations (1):
- Ankara University Medical School Anesthesiology and ICU Department, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Alibayli L, Cakar Turhan KS, Baytas V, Karadag Erkoc S, Bermede O, Kocaoglu H. Modified frailty index (mFI): is it a predictor for early postoperative complications in arthroplasty surgery? Eur Rev Med Pharmacol Sci. 2024 Feb;28(3):1002-1014. doi: 10.26355/eurrev_202402_35336. PMID 38375705